CLINICAL TRIAL: NCT06149338
Title: Vie Scope Versus Macintosh Laryngoscope in Expected Easy Airways: A Randomized Controlled Trial
Brief Title: The Rate of Successful Intubation and the Required Time for Intubation, Using Vie Scope and Macintosh Laryngoscope Will be Compared, in Order to Evaluate the Efficacy of Vie Scope in Comparison With Macintosh in Expected Easy Airways.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Andrew's General Hospital, Patras, Greece (Other)
Responsible Party: Principal Investigator, Vasileios Boviatsis, Principal Investigator, St. Andrew's General Hospital, Patras, Greece
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 141/09.07.2023
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Laryngoscopy
Keywords: Vie Scope; Macintosh; Rate of successful intubation; Intubation time

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients being intubated using Macintosh laryngoscope (Experimental)
  Interventions: Device: Macintosh laryngoscope
- Patients being intubated using Vie Scope laryngoscope (Experimental)
  Interventions: Device: Vie Scope

INTERVENTIONS:
Device: Macintosh laryngoscope — Macintosh laryngoscope has been the gold standard for endotracheal intubation since the middle of 20th century. During laryngoscopy and direct vision of the vocal cords, an endotracheal tube is passed into the trachea, establishing the airway.
  Arms: Patients being intubated using Macintosh laryngoscope
Device: Vie Scope — Vie Scope is a laryngoscope, whose function is relied on Seldinger technique. Firstly, bougie is passed through the translucent barrel of Vie Scope under direct vision between the vocal cords and into the trachea. Then, Vie Scope is removed and an endotracheal tube is passed over the bougie, which will be finally removed. The inflation of the endotracheal tube's cuff is followed by ventilation and confirmation of the tube placement.
  Arms: Patients being intubated using Vie Scope laryngoscope

SUMMARY:
The rate of successful intubation and the required time for intubation, using Vie Scope and Macintosh Laryngoscope will be compared, in order to evaluate the efficacy of Vie Scope in comparison with Macintosh in expected easy airways. Hence, a prospective randomized controlled single-blind superiority clinical trial will be conducted.

Inclusion criteria: patients of both sexes, positive or negative rapid test for COVID-19 or possible contamination, age ≥18 years old, BMI: 18.5 - 30 kg/m2, visualization of the glottis grade 1 or 2, according to Cormack-Lehane Classification.

Exclusion criteria: age under 18 years old, BMI under 18.5 kg/m2 and BMI over 30 kg/m2, visualization of the glottis grade 3 - 4, according to Cormack-Lehane Classification.

The laryngoscopy and intubation of the patients will be attempted by the same person-resident of Anesthesiology, under the supervision of experienced Anesthesiologist consultants.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Positive or negative rapid test for COVID-19 or possible contamination
* Age ≥18 years old
* BMI: 18.5 - 30 kg/m2
* Visualization of the glottis grade 1 or 2, according to Cormack-Lehane Classification.

Exclusion Criteria:

* Age under 18 years old
* BMI under 18.5 kg/m2 and BMI over 30 kg/m2
* Visualization of the glottis grade 3 - 4, according to Cormack-Lehane Classification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Andrew's General Hospital of Patras, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Being Intubated Using Macintosh Laryngoscope | Patients Being Intubated Using Vie Scope Laryngoscope
Started | 132 | 132
Completed | 132 | 132
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Being Intubated Using Macintosh Laryngoscope | Patients Being Intubated Using Vie Scope Laryngoscope | Total
Number analyzed (Participants) | 132 | 132 | 264
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63.5 [48 to 74.5] | 67 [53.5 to 75] | 65 [50.5 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 62 | 130
  Male | 64 | 70 | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 132 | 132 | 264
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Greece | 132 | 132 | 264

OUTCOME MEASURES:

1. Primary Outcome: Rate of Successful Intubation With One Attempt
Description: This outcome depends on whether the intubation of each patient will be successful or not, after the first attempt of intubation
Time Frame: Evaluation immediately after the first attempt of intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Being Intubated Using Macintosh Laryngoscope | Patients Being Intubated Using Vie Scope Laryngoscope
Number analyzed (Participants) | 132 | 132
Participants | 132 | 119
Statistical Analysis 1: Comparison: Patients Being Intubated Using Macintosh Laryngoscope vs Patients Being Intubated Using Vie Scope Laryngoscope; Test type: Superiority; p = 0.0002, Chi-squared — Threshold for statistical significance: p < 0.05
Statistical Analysis 2: Comparison: Patients Being Intubated Using Macintosh Laryngoscope vs Patients Being Intubated Using Vie Scope Laryngoscope; Test type: Superiority; p < 0.05, Fisher Exact

2. Primary Outcome: Mean Intubation Time
Description: Mean time interval required for intubation, which is determined from the time of the insertion of the laryngoscope into the patient's mouth until the time of the inflation of the tube's cuff on each patient
Time Frame: Assessment of the required mean time interval for intubation, immediately after the insertion of laryngoscope's blade into the patient's mouth
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Patients Being Intubated Using Macintosh Laryngoscope | Patients Being Intubated Using Vie Scope Laryngoscope
Number analyzed (Participants) | 132 | 132
seconds | 8.08 (5.34) | 16.65 (5.02)
Statistical Analysis 1: Comparison: Patients Being Intubated Using Macintosh Laryngoscope vs Patients Being Intubated Using Vie Scope Laryngoscope; Test type: Superiority; p < 0.0001, Kruskal-Wallis — Threshold for statistical significance: p < 0.05

3. Secondary Outcome: Rate of Successful Intubation
Description: This outcome depends on whether the intubation of each patient will be successful or not
Time Frame: Evaluation immediately after the intubation attempts
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Being Intubated Using Macintosh Laryngoscope | Patients Being Intubated Using Vie Scope Laryngoscope
Number analyzed (Participants) | 132 | 132
Participants | 132 | 124
Statistical Analysis 1: Comparison: Patients Being Intubated Using Macintosh Laryngoscope vs Patients Being Intubated Using Vie Scope Laryngoscope; Test type: Superiority; p = 0.0041, Chi-squared — Threshold for statistical significance: p < 0.05
Statistical Analysis 2: Comparison: Patients Being Intubated Using Macintosh Laryngoscope vs Patients Being Intubated Using Vie Scope Laryngoscope; Test type: Superiority; p < 0.05, Fisher Exact

4. Secondary Outcome: Visualization of the Glottis, According to Cormack Lehane Classification
Description: Ability to visualize the glottis, according to Cormack Lehane classification. The specific classification is divided into four grades (1-4). The higher the grade, the higher the likelihood of difficult intubation.
Time Frame: This outcome will be evaluated during laryngoscopy and intubation of each patient
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Being Intubated Using Macintosh Laryngoscope | Patients Being Intubated Using Vie Scope Laryngoscope
Number analyzed (Participants) | 132 | 132
Participants
  Grade 1 | 100 | 102
  Grade 2a | 20 | 21
  Grade 2b | 12 | 9
Statistical Analysis 1: Comparison: Patients Being Intubated Using Macintosh Laryngoscope vs Patients Being Intubated Using Vie Scope Laryngoscope; Test type: Superiority; p = 0.7895, Kruskal-Wallis — Threshold for statistical significance: p < 0.05

ADVERSE EVENTS:
Time Frame: During the intubation process (< 60 sec), the patient was simultaneously assessed for complications like injury of the structures of the upper airway, caused by the manipulations of the airway operator for the airway establishment. After the successful endotracheal intubation, the patients were not reassessed for any complications.
Arm/Group | Patients Being Intubated Using Macintosh Laryngoscope | Patients Being Intubated Using Vie Scope Laryngoscope
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/132
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/132
Other Adverse Events (participants affected / at risk) | 0/132 | 0/132

LIMITATIONS AND CAVEATS:
The airway operator was an anesthesiologist trainee with minimum experience. Thereby, the outcomes are not indicative of the Macintosh and Vie Scope use by consultants. Moreover, patients in both groups were not reassessed after endotracheal intubation, by direct laryngoscopy, in order to detect any potential complications. Finally, the current study was focused on the easy airway management of adults, providing no data about difficult airway management in adults and pediatric patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT06149338/Prot_SAP_001.pdf